CLINICAL TRIAL: NCT04645537
Title: Finnish AntiCoagulation in Atrial Fibrillation (FinACAF)
Acronym: FinACAF
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Aalto University (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Mika Lehto, Docent, MD, PhD, Cardiologist, Helsinki University Central Hospital
Other Study IDs: 70142
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Anticoagulation therapy; Warfarin; NOAC; DOAC; Novel oral anticoagulants; FinACAF; Finland; AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FinACAF cohort: The study cohort consists of all patients with AF diagnosis (ICD-10 I48) living in Finland during 1.1.2004-31.12.2018. The study cohort is obtained from data of Finnish national registries. Patients with permanent residence in Finland less than 12 months prior to index date are excluded from the study.

SUMMARY:
The aim of FINACAF study is to evaluate the incidence and risk of stroke, systemic thromboembolic events, myocardial infarction, major bleeding events, and mortality in relation to different attitudes regarding stroke prevention treatment among AF patients.

The study with cohort design is conducted as a nationwide retrospective register-based linkage study using data obtained from the Finnish health care registers.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia, its prevalence increases with age, and it presents with a wide spectrum of symptoms and severity. It has been estimated that number of AF patients is about 150 000 in Finland, and this number will be increased at least two-fold until year 2050.

The aim of this study is to evaluate the incidence and risk of stroke, systemic thromboembolic events, myocardial infarction, major bleeding events, and mortality in relation to different attitudes regarding stroke prevention treatment among AF patients.

An important part of the study is also the assessment of cost effectiveness of different OAC therapies. The risks mentioned above are separately evaluated with different management levels of warfarin therapy as well as with different NOACs and in patients without OAC treatment. The study population is also characterized according to co-morbidity, interactive medications and antiarhythmic drugs in use.

The study with cohort design is conducted as a nationwide retrospective register-based linkage study using data obtained from the Finnish health care registers. The study cohort consists of patients from six hospital district areas having a diagnosis of AF. The catchment population of these six districts is about 3.5 million; 64 % of the total Finnish population 5.5 million.

The study is register-based and patients will not be contacted in any phase of the study. Thus, no patient consents will be needed according to Finnish legislation. All patient data handled by the researchers will anonymous, ensuring full data protection of the patients.

ELIGIBILITY:
Inclusion Criteria:

Subject has an International Classification of Diseases (ICD-10 version 10) diagnosis code I48 for AF during 1.1.2004-31.12.2018 in any of the used registries

Exclusion Criteria:

* No ICD-10 I48 diagnose in any of the study registries.
* Subjects with age below 18 years at index date
* Patients with permanent residence in Finland less than 12 months prior to index date.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all AF patients of the study region (Six pre-selected hospital districts with laboratory data available) during 1.1.2004-31.06.2018, including newly diagnosed patients with ICD-10 I48 diagnose code.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Follow-up period 1/2004-12/2018
  All-cause, stroke, myocardial infarction,systemic thromboembolic events, bleeding events
Bleeding events | Follow-up period 1/2004-12/2018
  Intracranial hemorrage, Gastrointestinal hemorrage, other major bleeding events
Ischemic Stroke | Follow-up period 1/2004-12/2018
  ICD-10: I63, I64, I693-I698, G45
Myocardial infarction | Follow-up period 1/2004-12/2018
  ICD-10: I21, I22
Systemic Thromboembolism | Follow-up period 1/2004-12/2018
  Other than stroke or myocardial infarction

SECONDARY OUTCOMES:
Anemia | Follow-up period 1/2004-12/2018
  Decrement of haemoglobin during follow-up period. Detailed description available in Statistical Analysis plan under secondary objectives.
Renal failure | Follow-up period 1/2004-12/2018
  Time to renal impairment is defined as the time from index date to time when serum creatinine level is under the reference value.
Dementia | 1/2004-12/2018
  Time to dementia diagnosis in patients without pre-existing dementia, ICD: F00,F01, F02, F03
Healthcare Service costs | 1/2004-12/2018
  The Diagnosis-Related Groups (DRG) are based on the Finnish version of the Nordic Classification of Surgical Procedures codes for diagnostic and treatment procedures, and the respective Nordic Diagnosis-Related Groups patient classifications. Respectively, the patient-level data for primary care (with diagnosis and activity information) are grouped using the Ambulatory and Primary Care-Related Patient Groups (APR) grouper, a grouping system equivalent to DRG used in hospital care.
  The detailed description available in Statistical Analysis plan under secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Mika Lehto, MD,PhD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lehtonen O, Halminen O, Airaksinen KEJ, Haukka J, Putaala J, Mustonen P, Teppo K, Kouki E, Aro AL, Hartikainen J, Lehto M, Linna M. Cost Differences Between Oral Anticoagulation Therapies in Patients with Atrial Fibrillation in Finland. Drugs Real World Outcomes. 2025 Dec;12(4):631-641. doi: 10.1007/s40801-025-00519-5. Epub 2025 Oct 7. PMID 41057675
- [Derived] Lehto J, Bjorn R, Halminen O, Linna M, Haukka J, Putaala J, Mustonen P, Kinnunen J, Hartikainen J, Airaksinen JKE, Kiviniemi TO, Lehto M. Quality of anticoagulation and outcomes after mechanical aortic valve replacement in patients with atrial fibrillation: a nationwide cohort study. Eur Heart J Qual Care Clin Outcomes. 2025 Aug 11;11(5):654-664. doi: 10.1093/ehjqcco/qcaf028. PMID 40366898
- [Derived] Teppo K, Airaksinen KEJ, Biancari F, Jaakkola J, Halminen O, Linna M, Haukka J, Putaala J, Mustonen P, Kinnunen J, Luojus A, Hartikainen J, Aro AL, Lehto M. Aortic Stenosis and Outcomes in Patients With Atrial Fibrillation: A Nationwide Cohort Study. J Am Heart Assoc. 2023 May 2;12(9):e029337. doi: 10.1161/JAHA.122.029337. Epub 2023 Apr 29. PMID 37119067
- [Derived] Lehto M, Haukka J, Aro A, Halminen O, Putaala J, Linna M, Mustonen P, Kinnunen J, Kouki E, Niiranen J, Luojus A, Tiili P, Itainen-Stromberg S, Hartikainen J, Airaksinen JKE; FinACAF study group. Comprehensive nationwide incidence and prevalence trends of atrial fibrillation in Finland. Open Heart. 2022 Nov;9(2):e002140. doi: 10.1136/openhrt-2022-002140. PMID 36414332
- [Derived] Teppo K, Jaakkola J, Biancari F, Halminen O, Putaala J, Mustonen P, Haukka J, Linna M, Kinnunen J, Luojus A, Itainen-Stromberg S, Penttila T, Niemi M, Hartikainen J, Airaksinen KJ, Lehto M. Mental health conditions and use of rhythm control therapies in patients with atrial fibrillation: a nationwide cohort study. BMJ Open. 2022 Aug 30;12(8):e059759. doi: 10.1136/bmjopen-2021-059759. PMID 36041755
- [Derived] Biancari F, Teppo K, Jaakkola J, Halminen O, Linna M, Haukka J, Putaala J, Mustonen P, Kinnunen J, Hartikainen J, Aro A, Airaksinen J, Lehto M. Income and outcomes of patients with incident atrial fibrillation. J Epidemiol Community Health. 2022 Jun 15;76(8):736-42. doi: 10.1136/jech-2022-219190. Online ahead of print. PMID 35705362
- [Derived] Teppo K, Jaakkola J, Airaksinen KEJ, Biancari F, Halminen O, Putaala J, Mustonen P, Haukka J, Hartikainen J, Luojus A, Niemi M, Linna M, Lehto M. Mental Health Conditions and Nonpersistence of Direct Oral Anticoagulant Use in Patients With Incident Atrial Fibrillation: A Nationwide Cohort Study. J Am Heart Assoc. 2022 Mar 15;11(6):e024119. doi: 10.1161/JAHA.121.024119. Epub 2022 Mar 1. PMID 35229612

DOCUMENTS (1):
  • Study Protocol (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04645537/Prot_001.pdf